CLINICAL TRIAL: NCT00733824
Title: A Phase I/II Study of Intravenous AMD3100 Added to a Mobilization Regimen of G-CSF to Increase the Number of Autologous Peripheral Blood Stem Cells Collected From Patients With Lymphoma
Brief Title: Intravenous AMD3100 for Collection of Autologous Peripheral Blood Stem Cells in Patients With Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0897 / 201105349
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Plerixafor; Lymphoma; Hematopoietic Stem Cell Mobilization; Transplantation, Autologous; Receptors, CXCR4
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — plerixafor; Granulocyte Colony-Stimulating Factor; Filgrastim; Blood Component Removal; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  160 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  Interventions: Drug: AMD3100; Drug: G-CSF; Procedure: Apheresis
- Cohort 2 (Experimental): 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  240 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  Interventions: Drug: AMD3100; Drug: G-CSF; Procedure: Apheresis
- Cohort 3 (Experimental): 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  320 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  Interventions: Drug: AMD3100; Drug: G-CSF; Procedure: Apheresis
- Cohort 4 (Experimental): 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  400 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  Interventions: Drug: AMD3100; Drug: G-CSF; Procedure: Apheresis
- Phase II (Experimental): 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  MTD as determined in Phase I IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  Interventions: Drug: AMD3100; Drug: G-CSF; Procedure: Apheresis

INTERVENTIONS:
Drug: AMD3100
  Other Names: Plerixafor
Drug: G-CSF
  Other Names: Neupogen; Filgrastim
Procedure: Apheresis
  Other Names: Leukopheresis

SUMMARY:
This study will evaluate the safety and efficacy of intravenous AMD3100 added to a standard G-CSF mobilization regimen of patients undergoing autologous stem cell transplantation for lymphoma.

The investigators hypothesize that after stem cell mobilization with G-CSF plus IV AMD3100, a significantly higher proportion of lymphoma patients will collect ≥ 2 x 10E6 CD34+ cells/kg.

DETAILED DESCRIPTION:
Autologous stem cell transplantation (ASCT) is indicated for patients with non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL) who have primary progressive disease or who relapse after a chemotherapy-induced complete remission. For these patients, as for other patients undergoing autologous transplantation, the number of CD34+ cells collected is a reliable predictor of neutrophil and platelet (PLT) engraftment after transplantation.

AMD3100 (plerixafor) is a promising new mobilizing agent that has demonstrated efficacy in patients with NHL, HL, and multiple myeloma (MM). Although efficacious, the subcutaneous dosing of AMD3100 requires that patients receive the drug in the evening prior to apheresis, which can present logistical problems. Intravenous dosing of AMD3100 may result in a faster rise in peripheral CD34+ cell count, so that the drug can be administered the same day as apheresis. Intravenous dosing may also increase the peak CD34+ cell count, improving the number of CD34+ cells collected via apheresis.

This Phase I/II study will evaluate the safety and efficacy of intravenous AMD3100 added to the standard G-CSF mobilization regimen of patients undergoing autologous stem cell transplantation for Hodgkin and non-Hodgkin lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Diagnosis of HL or NHL eligible for autologous transplantation
* 30 days since last cycle of chemotherapy
* ECOG performance status of 0 or 1
* The patient has recovered from all acute toxic effects of prior chemotherapy
* WBC >3.0 X 109/l
* Absolute PMN count >1.5 X 109/l
* PLT count >100 X 109/l
* Serum creatinine ≤ 2.2 mg/dl
* AST (SGOT), ALT (SGPT) and total bilirubin < 2X upper limit of normal (ULN)
* Left ventricle ejection fraction > 45% (by ECHO or MUGA scan)
* FEV1 > 60% of predicted or DLCO > 45% of predicted
* Negative for HIV on standard transplant workup
* Signed informed consent
* Are surgically or biologically sterile or willing to practice acceptable birth control, as follows:

  * Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Women of child bearing potential must have a negative serum or urine pregnancy test at the time of enrollment. Acceptable methods of birth control include oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives and abstinence.
  * Males must agree to abstain from sexual activity or agree to utilize a medically approved contraception method during and for 3 months after the treatment period

Exclusion Criteria:

* A co-morbid condition which, in the view of the investigator, renders the patient at high risk for treatment complications
* Patients who have failed previous collections
* A residual acute medical condition resulting from prior chemotherapy
* Acute infection
* Fever (temp >38C/100.4F) on the day of start of treatment
* Positive pregnancy test in female patients
* Lactating females
* Patients of child bearing potential unwilling to implement adequate birth control
* Patients whose actual body weight exceeds 150% of their ideal body weight
* History of ventricular arrhythmias
* Patients who previously received experimental therapy within 4 weeks of enrolling in this study or who are currently enrolled in another experimental study during the mobilization phase
* Patients who have deterioration of their clinical status or laboratory parameters between the time of enrollment and transplantation such that they no longer meet entry criteria may be removed from study at the discretion of the treating physician, principal investigator, or sponsor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda F. Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devine SM, Flomenberg N, Vesole DH, Liesveld J, Weisdorf D, Badel K, Calandra G, DiPersio JF. Rapid mobilization of CD34+ cells following administration of the CXCR4 antagonist AMD3100 to patients with multiple myeloma and non-Hodgkin's lymphoma. J Clin Oncol. 2004 Mar 15;22(6):1095-102. doi: 10.1200/JCO.2004.07.131. PMID 15020611
- [Background] Flomenberg N, Devine SM, Dipersio JF, Liesveld JL, McCarty JM, Rowley SD, Vesole DH, Badel K, Calandra G. The use of AMD3100 plus G-CSF for autologous hematopoietic progenitor cell mobilization is superior to G-CSF alone. Blood. 2005 Sep 1;106(5):1867-74. doi: 10.1182/blood-2005-02-0468. Epub 2005 May 12. PMID 15890685
- [Background] DiPersio JF, Micallef I, Stiff PJ, et al. A Phase III, Multicenter, Randomized, Double-Blind, Placebo Controlled, Comparative Trial of AMD3100 (Plerixafor)+G-CSF vs. Placebo+G-CSF in Non-Hodgkin's Lymphoma (NHL) Patients for Autologous Hematopoietic Stem Cell (aHSC) Transplantation. ASH Annual Meeting Abstracts. November 16, 2007 2007;110(11):601-.
- [Background] Cashen A, Lopez S, Gao F, Calandra G, MacFarland R, Badel K, DiPersio J. A phase II study of plerixafor (AMD3100) plus G-CSF for autologous hematopoietic progenitor cell mobilization in patients with Hodgkin lymphoma. Biol Blood Marrow Transplant. 2008 Nov;14(11):1253-61. doi: 10.1016/j.bbmt.2008.08.011. PMID 18940680
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Cohort 1: * 240 µg/kg SC AMD3100 Day -5
  * 10 µg/kg SC G-CSF Day -4 thru Day -1
  * 160 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  * Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
- Phase I - Cohort 2: * 240 µg/kg SC AMD3100 Day -5
  * 10 µg/kg SC G-CSF Day -4 thru Day -1
  * 240 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  * Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
- Phase I - Cohort 3: * 240 µg/kg SC AMD3100 Day -5
  * 10 µg/kg SC G-CSF Day -4 thru Day -1
  * 320 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  * Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
- Phase I - Cohort 4: 240 µg/kg SC AMD3100 Day -5 10 µg/kg SC G-CSF Day -4 thru Day -1 400 µg/kg IV AMD3100 and 10 µg/kg SC G-CSF Day 1 Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
- Phase II: * 240 µg/kg SC AMD3100 Day -5
  * 10 µg/kg SC G-CSF Day -4 thru Day -1
  * MTD as determined in Phase I IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  * Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
Period: Phase I
Arm/Group | Phase I - Cohort 1 | Phase I - Cohort 2 | Phase I - Cohort 3 | Phase I - Cohort 4 | Phase II
Started | 10 | 3 | 6 | 6 | 0
Completed | 9 | 3 | 6 | 6 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I - Cohort 1 | Phase I - Cohort 2 | Phase I - Cohort 3 | Phase I - Cohort 4 | Phase II
Started | 0 | 0 | 0 | 0 | 36
Completed | 0 | 0 | 0 | 0 | 36
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II | Total
Number analyzed (Participants) | 10 | 3 | 6 | 6 | 36 | 61
Age, Continuous [Median (Full Range); unit: years] | 49.5 [24 to 69] | 48 [30 to 50] | 50 [25 to 53] | 47 [25 to 59] | 60 [23 to 73] | 53 [23 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 2 | 12 | 20
  Male | 7 | 2 | 4 | 4 | 24 | 41
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 6 | 6 | 36 | 61

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of IV AMD3100 + G-CSF in Mobilization of Peripheral Blood Stem Cell in Patients With Lymphoma (Phase I Only)
Description: * MTD: the highest dose level of AMD3100 at which ≤ 1 of 6 participants experience a dose limiting toxicity (DLT). The MTD will be the Phase II dose.
  * DLT: selected grade III or higher (hematologic, cardiac, pulmonary, hepatobiliary/pancreatic, renal, or CNS) not attributable to any other cause.
Time Frame: 7 days from first dose of IV AMD3100
Measure: Number; unit: micrograms/kilograms
Arm/Group | Phase 1 (Dose Levels 1-4)
Number analyzed (Participants) | 25
micrograms/kilograms | 400

2. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities in Phase I Portion of Study
Description: Dose limiting toxicity: selected grade III or higher (hematologic, cardiac, pulmonary, hepatobiliary/pancreatic, renal, or CNS) not attributable to any other cause.
Time Frame: 7 days from first dose of IV AMD3100
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 10 | 3 | 6 | 6
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Kinetics of Stem Cell Mobilization Using IV AMD3100 as Measured by Median Fold Change in the Number of CD34+ Cells After AMD3100 IV Administration
Time Frame: From baseline to Day 1
Measure: Median (Full Range); unit: fold change
Arm/Group | Phase 1 and Phase 2 Participants
Number analyzed (Participants) | 61
fold change | 2.1 [0.8 to 7.0]

4. Secondary Outcome: Pharmacodynamic Response to a Dose of SC AMD3100 as Measured by Mean Percentage of the Circulating CD34+ Count With the 34+RA-123+/- Phenotype
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mean percentage of total CD34+ cells
Arm/Group | Phase 1 and Phase 2 Participants
Number analyzed (Participants) | 25
mean percentage of total CD34+ cells | 49.0 (13.2)

5. Secondary Outcome: Toxicity of the Combination IV AMD3100 and G-CSF to Mobilize ≥ 2 x 106 CD34+ Cells/kg as Measured by Number of Participants Who Experience Grade 3 or Higher Adverse Event Broken Down by Adverse Event
Time Frame: 30 days post transplant
Measure: Number; unit: participants
Groups:
- Phase II: 240 µg/kg SC AMD3100 Day -5
  10 µg/kg SC G-CSF Day -4 thru Day -1
  MTD as determined in Phase I IV AMD3100 and 10 µg/kg SC G-CSF Day 1
  Pheresis (this will be repeated on Day 2 through Day 4 until target of ≥5X106 CD34+ cell/kg is reached)
  AMD3100
  G-CSF
  Apheresis
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II
Number analyzed (Participants) | 10 | 3 | 6 | 6 | 36
participants
  Hemoglobin | 3 | 2 | 4 | 4 | 20
  Leukocytes (WBC) | 4 | 3 | 6 | 6 | 32
  Lymphopenia | 3 | 3 | 3 | 5 | 29
  Neutrophils (ANC) | 3 | 3 | 6 | 6 | 29
  Platelets | 5 | 3 | 5 | 6 | 34
  Alkaline phosphtase | 1 | 0 | 0 | 0 | 0
  SGPT (ALT) | 1 | 0 | 1 | 0 | 0
  Hypoxia | 3 | 0 | 0 | 0 | 0
  Hypotension | 0 | 1 | 0 | 0 | 2
  Mucositis | 0 | 0 | 0 | 1 | 0
  Infection with neutropenia | 0 | 0 | 0 | 2 | 0
  Febrile neutropenia | 0 | 0 | 0 | 4 | 0
  INR | 0 | 0 | 0 | 1 | 0
  PTT | 0 | 0 | 0 | 1 | 8
  Bleeding at catheter site | 0 | 0 | 0 | 0 | 1
  Hemorrhage - spleen | 0 | 0 | 0 | 0 | 1
  Atrial fibrillation | 0 | 0 | 0 | 0 | 1
  Diarrhea | 0 | 0 | 0 | 0 | 1
  Ileus | 0 | 0 | 0 | 0 | 1
  Nausea | 0 | 0 | 0 | 0 | 1
  Vomiting | 0 | 0 | 0 | 0 | 1
  Hyperbilirubinemia | 1 | 0 | 0 | 0 | 2
  Fungal infection | 0 | 0 | 0 | 0 | 1
  Opportunistic infection | 0 | 0 | 0 | 0 | 1
  Clostridium difficile | 0 | 0 | 0 | 0 | 1
  Colitis | 0 | 0 | 0 | 0 | 1
  E. coli infection | 0 | 0 | 0 | 0 | 1
  Leptotrichia | 0 | 0 | 0 | 0 | 1
  Lung infection (pneumonia) | 0 | 0 | 0 | 0 | 1
  Staph infection | 0 | 0 | 0 | 0 | 1
  Typhlitis | 0 | 0 | 0 | 0 | 1
  Glucose - high | 0 | 0 | 0 | 0 | 2
  Magnesium - high | 0 | 0 | 0 | 0 | 1
  Potassium - low | 1 | 0 | 0 | 2 | 1
  Sodium - low | 0 | 0 | 0 | 1 | 6
  Cough | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/3 | 0/6 | 0/6 | 2/36
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3 | 6/6 | 6/6 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=6) | Phase II (N=36)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Death - disease progression (General disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhage - spleen (General disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=6) | Phase II (N=36)
Abdominal distension/bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 2 | 2 | 3
Albumin - low (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 2
Alkaline phosphatase (Investigations) | 7 | 1 | 5 | 6 | 26
Allergic reaction (platelets) (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (joint) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 7
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 7
Bleeding at catheter site (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 14
Calcium (high) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Calcium - low (Metabolism and nutrition disorders) | 2 | 0 | 1 | 6 | 4
Catheter site - neck pain (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 1 | 4
Chest (tightness, pressure) (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Clostridium difficile (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 1
Creatinine (Investigations) | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Diaphoresis (General disorders) | 1 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 0 | 1 | 6 | 18
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
E. coli infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 0 | 0 | 5
Fatigue (General disorders) | 8 | 3 | 2 | 5 | 8
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 4 | 0
Fever (General disorders) | 1 | 0 | 0 | 0 | 0
Flu-like syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
General body ache (General disorders) | 0 | 0 | 1 | 0 | 0
Glucose - high (Metabolism and nutrition disorders) | 4 | 0 | 0 | 3 | 3
Glucose - low (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
HSV blister - lip (General disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 1 | 1 | 4
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 9 | 2 | 6 | 6 | 27
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinemia (Investigations) | 1 | 0 | 0 | 1 | 3
Hypersalivation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 0 | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
INR (Investigations) | 0 | 0 | 0 | 3 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Infection with neutropenia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Leptotrichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Leukocytes (WBC) (Investigations) | 6 | 3 | 6 | 6 | 33
Lung infection (pneumonia) (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymphopenia (Investigations) | 6 | 3 | 3 | 5 | 31
Magnesium (high) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Magnesium - low (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1
Mucositis (Gastrointestinal disorders) | 5 | 0 | 0 | 1 | 0
Muscle cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Muscle weakness - left arm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 4 | 4 | 13
Neutrophils (ANC) (Investigations) | 3 | 3 | 6 | 6 | 29
Night sweats (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Opportunistic infection w/grade 2 or higher lymphopenia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
PTT (Investigations) | 0 | 0 | 0 | 4 | 15
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Platelets (Investigations) | 7 | 0 | 5 | 6 | 35
Potassium - low (Metabolism and nutrition disorders) | 3 | 0 | 0 | 4 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Rigors/chills (General disorders) | 0 | 0 | 0 | 0 | 1
SGOT (AST) (Investigations) | 3 | 0 | 1 | 4 | 6
SGPT (ALT) (Investigations) | 6 | 0 | 2 | 5 | 5
Sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 16
Sinus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0
Sodium - low (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 6
Staph infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Typhlitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Uric acid (high) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 1 | 2 | 5
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0 | 0
Whole body pain (General disorders) | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes